CLINICAL TRIAL: NCT05898061
Title: Optimal Lidocaine Propofol Mixture for Painless Induction of Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fawzy Abbas Badawy, Optimal lidocaine propofol mixture for painless induction of anesthesia, Sohag University
Other Study IDs: Soh-Med-22-11-15
Record Dates: First submitted 2023-04-30; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Pain, During Injection of Propofol for Induction of Anesthesia
Keywords: Propofol - Lidocaine - Painless Induction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research will be carried out in order to determine the optimal lidocaine dose in propofol lidocaine mixture to prevent pain on propofol injection during induction of general anesthesia using a modified Dixon's up-and-down method. Patients & methods: Include assessment of severity of pain on propofol injection using seven doses of lidocaine in lidocaine propofol mixture in ASA I&II patients aged 18-60 years with exclusion of patients with history of drug allergy, hepatic or renal impairment, cardiac problems, neurologic deficits or psychiatric disorders.

The primary outcome will be pain scale during injection and volume of propofol-lidocaine mixture used. Secondary outcome will be increase in heart rate and/or hand or forearm withdrawal during injection, patient satisfaction, demographic data, type and duration of surgery, Time for unconsciousness.

Aim of the work: To determine the Minimal effective dose of lidocaine in propofol lidocaine mixture to achieve painless induction of anesthesia using propofol.

DETAILED DESCRIPTION:
Rapid onset of action, smooth induction, favorable recovery and low rate of adverse effects have made propofol the most commonly used intravenous anesthetic for induction and maintenance of anesthesia. However, pain associated with propofol injection is still considered by many patients as the worst prioperative unpleasant experience.1 Therefore, a diversity of techniques have been suggested in the literature to solve this problem including pretreatment with local anesthetics, opiates, ketamine and alfentanil. 2-5 New propofol formulation was another way to alleviate this pain.6 Among these techniques lidocaine was investigated extensively whether as a pretreatment with the use of tourniquet, which is a time consuming technique, or mixed with propofol. Evaluation of optimal dose of lidocaine in propofol lidocaine mixture was widely assessed. However, evaluation of optimal lidocaine dose in propofol lidocaine mixture to prevent pain with newer formulations of propofol should be further evaluated. We hypothesize that optimal dose of lidocaine to alleviate pain with propofol injection might need further evaluation.

Patients and methods

This prospective randomized and double blinded study will be conducted in Sohag University Hospital after obtaining approval from Institutional Review Board and written informed consent from all patients before enrolment in this study. Patients scheduled for elective surgery under general anesthesia, aged 18 to 60 years and American Society of Anesthesiologists (ASA)physical status I & II will be selected for this study. Patients with history of drug allergy, hepatic or renal impairment, cardiac problems, neurologic deficits, psychiatric disorders or anxious patients who need sedation preoperatively will be excluded from the study.

Before entering the operating room premedication will not be allowed. In the operating room 20 gauge cannula will be inserted into a vein on the dorsum of the non-dominant hand & basic monitoring (pulse oximetry, electrocardiography, noninvasive blood pressure & end tidal carbon dioxide) will be applied to the patient before induction and throughout the procedure.

Mixtures of propofol, lidocaine and saline will be prepared by an anesthetist who is not involved in the study team according to the lidocaine dose sequence as shown in table (1) resulting into eight mixtures. The mixture will be injected at a rate of 20ml/minute using syringe pump until patient loose consciousness. The anesthetist who inject the propofol and the patient will be blinded to the lidocaine dose in the mixture.

Table 1 propofol lidocaine mixtures Mixture Propofol Lidocaine 2% (ml)(20mg/ml) Lidocaine concentration (%)

1. 20ml 0.5
2. 20ml 1 0.095
3. 20ml 1.5 0.139
4. 20ml 2 0.181
5. 20ml 2.5 0.222
6. 20ml 3 0.26
7. 20ml 3.5 0.297
8. 20ml 4 0.333

Pain scale will be explained to all patients preoperatively and they will be asked to report for pain sensation (no pain or mild, moderate or severe pain) The dose of lidocaine, in propofol lidocaine mixture, administered to each patient will be determined by the response of the previous patient using a modified Dixon's up-and-down method (using 10mg as a step size). The first patient will receive a mixture with 10mg lidocaine. If the patient report pain with propofol injection, then the next patient will receive a mixture with 10mg higher dose of lidocaine, if the patient report no pain with injection, then the next patient will receive a mixture with 10mg lower dose of lidocaine. The study will continue until we obtain seven crossover midpoints (No limited number).

The minimal effective dose of lidocaine that results in painless injection of propofol for 50% (ED50) of patients will be determined by calculating the midpoint dose of all independent pairs of patients after at least seven crossover points.

The following data will be recorded; Primary outcome: pain scale during injection and volume of propofol-lidocaine mixture used.

Secondary outcome: increase in heart rate and/or hand or forearm withdrawal during injection, patient satisfaction(will be assessed in the post anesthesia care unit (PACU) after regaining consciousness), demographic data, type and duration of surgery, Time for unconsciousness.

Aim of the work To determine the Minimal effective dose of lidocaine in propofol lidocaine mixture to achieve painless induction of anesthesia using propofol.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery under general anesthesia.
* Aged 18 to 60 years
* American Society of Anesthesiologists physical status I & II

Exclusion Criteria

* History of drug allergy
* Hepatic or renal impairment .Cardiac disease
* Neurologic deficits ,psychiatric disorders
* Anxious patients who need sedation preoperatively

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients scheduled for elective surgery under general anesthesia, aged 18 to 60 years and American Society of Anesthesiologists physical status I & II will be selected for this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain scale | 9 months
  Pain scale (mild, moderate or severe) during injection of propofol

SECONDARY OUTCOMES:
Heart rate | Before injection of propofol-lidocaine mixture and every minute for three minutes after start of injection
  Heart rate
time for unconsciousness | 2 minutes after start of injection of propofol
  time in seconds starting from injection of Propofol-lidocaine mixture until patient loose consciousness
patient satisfaction | 30 minutes after recovery
  describes satisfaction level of the patient regarding relief of propofol injection (not satisfied, less satisfied, satisfied, highly satisfied)
hand or forearm withdrawal | 2 minutes duration during injection of propofol
  withdrawal due to pain during injection of propofol

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Lembert N, Wodey E, Geslot D, Ecoffey C. [Prevention of pain on injection with propofol in children: comparison of nitrous oxide with lidocaine]. Ann Fr Anesth Reanim. 2002 Apr;21(4):263-70. doi: 10.1016/s0750-7658(02)00588-9. French. PMID 12033094
- [Background] Zahedi H, Nikooseresht M, Seifrabie M. Prevention of propofol injection pain with small-dose ketamine. Middle East J Anaesthesiol. 2009 Oct;20(3):401-4. PMID 19950734
- [Background] Iyilikci L, Balkan BK, Gokel E, Gunerli A, Ellidokuz H. The effects of alfentanil or remifentanil pretreatment on propofol injection pain. J Clin Anesth. 2004 Nov;16(7):499-502. doi: 10.1016/j.jclinane.2004.01.005. PMID 15590252
- [Background] Kobayashi Y, Naganuma R, Seki S, Aketa K, Ichimiya T, Namiki A. [Reduction of pain on injection of propofol: a comparison of fentanyl with lidocaine]. Masui. 1998 Aug;47(8):963-7. Japanese. PMID 9753961